CLINICAL TRIAL: NCT02752867
Title: Functional Magnetic Resonance Imaging Study to Explore the Mechanism and the Efficacy and Safety of Jianpi Yishen Huatan Granule for Cognitive Impairment After Acute Cerebral Infarction
Brief Title: An fMRI Study of Jianpi Yishen Huatan Granules for Cognitive Impairment After Acute Cerebral Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yunling Zhang, President of Dongfang Hospital, Dongfang Hospital Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140700108b
Record Dates: First submitted 2016-03-20; First posted 2016-04-27 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cognitive Impairment
Keywords: traditional Chinese medicine granules; Cognitive Impairment; Acute cerebral infraction; treatment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jianpi Yishen Huatan Granules group (Experimental): Treat with the prescription of Jianpi Yishen Huatan Granules and conventional treatment of ischemic stroke.
  Interventions: Drug: Jianpi Yishen Huatan Granules
- The control group (Placebo Comparator): Treat with the placebo which contain 5% of prescription of Jian Pi Yi Shen Hua Tan Granules and 95% dextrin and conventional treatment of ischemic stroke.
  Interventions: Other: the placebo

INTERVENTIONS:
Drug: Jianpi Yishen Huatan Granules — Jianpi Yishen Huatan Granules contain Herba cistanche，Fructus Alpinia Oxyphyllae，Rhodiola rosea, Polygala tenuifolia willd and Coptis chinensis.Jianpi Yishen Huatan Granules dissolved in water of 100 ml ,po, bid of each 90-days cycle. Number of treatment cycles: one
  Other Names: Jianpi Yishen Huatan Granules group
  Arms: Jianpi Yishen Huatan Granules group
Other: the placebo — Treat with the placebo which contain 5% of prescription of Jian Pi Yi Shen Hua Tan Granules and 95% dextrin.The placebo dissolved in water of 100 ml ,po, bid of each 90-days cycle. Number of cycles: one
  Other Names: the placebo group
  Arms: The control group

SUMMARY:
The purpose of this study is to explore the pathogenesis of cognitive impairment after acute cerebral infarction by applying the multimodal function MRI to dynamically observe the changes of the value of NAA,Cho,Cr,FA in a certain region in the brain and the function of the brain ,and to provide a visual instrument for evaluating the therapeutical effects of Chinese medicine through the application of multimodal function MRI to observe the changes of the neurotransmitter in certain area in the brain before and after the treatment.

DETAILED DESCRIPTION:
The present study is designed to assess the efficacy and safety of Jianpi Yishen Huatan granules with cognitive impairment after Acute Cerebral Infarction by fMRI and neuropsychology scales,as well as observe the symptoms,syndrome characteristics and neuropsychological changes of patients with cognitive dysfunction after acute cerebral infarction.And explore the pathogenesis of cognitive impairment after acute cerebral infarction by applying the multimodal function MRI to dynamically observe the changes of the value of NAA,Cho,Cr,FA in a certain region in the brain and the function of the brain ,and to provide a visual instrument for evaluating the therapeutical effects of Chinese medicine through the application of multimodal function MRI to observe the changes of the neurotransmitter in certain area in the brain before and after the treatment.

The sample size is 40 of which 20 are from the intervention group and 20 are from the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients conform to the diagnostic criteria of acute ischemic stroke.
* The cerebral infarction area lies in the blood supply area of middle cerebral artery: basal ganglia,corona radiate region or other subcortical regions..
* The cumulative infarction area is no more than 3.0 cm.
* Stroke onset within 21 days
* Age from forty to eighty, gender not limited
* Neuropsychological assessments: Montreal Cognitive Assessment Scale scores less than 26 points or MMSE scores range from 19 points to 26 points in literates or MMSE scores range from 17 points to 24 points in illiterates
* Informed and signed the informed consent

Exclusion Criteria:

* Transient Ischemic Attack
* Stroke patients with the causes of cerebral hemorrhage, subarachnoid hemorrhage, brain tumors, brain injury, or blood diseases and so on.
* Stroke with an onset of more than 21 days
* Cerebral embolism caused by atrial fibrillation resulted from rheumatic heart disease, coronary heart disease and other heart diseases.
* Patients who cannot cooperate with the check due to serious visual, hearing dysfunction, apraxia, aphasia.
* Patients with other neurological diseases which can affect cognitive function (for example:Alzheimer's Disease，Parkinson's disease, frontotemporal dementia，Huntington's disease)
* Patients with communication difficulties, or psychiatric disease
* Depression (Hamilton Depression Scale scores more than or equal to 17 points)
* Diagnosed with alcohol or drug dependence within the past six months
* With other diseases which can cause cognitive dysfunction, Such as trauma，tumor or infection of the central nervous system, metabolic disorders, normal pressure hydrocephalus , folic acid or vitamin B12 Deficiency, thyroid hypofunction,sever anemia,sever Parkinson's Disease, encephalitis, syphilis or HIV
* With a previous history of stroke and serious sequelae, and cannot cope with neuropsychological examination
* With severe primary diseases, and cannot comply with the above scheme

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Changes of the fMRI outcome after the treatment | 90 days
  Using the fMRI to measure the changes of neurotransmitter and brain function in the brain before and after the treatment.
Mini-mental state examination(MMSE) | 90 days
  MMSE is an acknowledged scale to measure cognition function from the aspects of orientation ability, memory, attention, calculation ability, recall and language,etc.
Montreal Cognitive Assessment scale(MoCA) | 90 days
  Using this scale to measure cognitive function
Stroop Color- Word Association Test（Stroop test） | 90 days
  This is a test used to find out the memory and executive function of patients.The test contains three small test.
Numerical sequence test（DS-S) | 90 days
  Using Numerical sequence test（DS-S) to examine memory
Digital color connection test (CCT) | 90 days
  Using Digital color connection test (CCT) to examine executive function and attention
Verbal memory test(HVLT) | 90 days
  Using Verbal memory test(HVLT) to examine verbal memory
Clinical Dementia Rating scale(CDR) | 90 days
  Using Clinical Dementia Rating scale(CDR) to measure the severity of dementia

SECONDARY OUTCOMES:
National institute of health stroke scale | 90 days
  Using National institute of health stroke scale to measure the severity of stroke
Modified Rankin scale | 90 days
  Using Modified Rankin scale to measure the recovery of neurological function
Activity of Daily Living Scale | 90 days
  Using this scale to measure daily living ability
Scores of Chinese medicine symptoms | 90 days
  Scores of Chinese medicine symptoms, which is a scale resulted from literature research, the argumentation of experts and clinical observation,contain 23 items of the core symptoms of cognitive impairment. And the scale is used to measure the changes of symptoms of Chinese medicine before and after treatment.

OTHER OUTCOMES:
whole blood cell test | 90 days
  blood routine test
routine urine test | 90 days
  routine urine test
Liver function | 90 days
  test the blood to detect the liver function,such as alanine aminotransferase(ALT) ,aspartate aminotransferase(AST),total bilirubin (TBIL), γ-glutamyl transferase(γ-GT).
electrocardiogram | 90 days
  electrocardiograms are given before the experiment and on the 90th day of the experiment to test the condition of the patients' heart.
homocysteine | 90 days
  detect the homocysteine in the blood
routine stool test | 90 days
  examine stool of the patients
kidney function | 90 days
  test the blood to detect the kidney function,such as blood urea nitrogen(BUN),creatinine (CRE),Uric acid(UA)

CONTACTS AND LOCATIONS:
Overall Officials: Yunling Zhang, Study Chair — Dongfang Hospital Beijing University of Chinese Medicine
Locations (1):
- Department of Neurology,Dongfang Hospital,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No